CLINICAL TRIAL: NCT01479842
Title: A Phase I, Dose-escalation Trial of Rituxan and Bendamustine in Combination With Bruton's Tyrosine Kinase Inhibitor, PCI-32765, in Patients With Relapsed Diffuse Large B-cell Lymphoma, Mantle Cell Lymphoma, or Indolent Non-Hodgkin's Lymphoma
Brief Title: Rituxan/Bendamustine/PCI-32765 in Relapsed DLBCL, MCL, or Indolent Non-Hodgkin's Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kami Maddocks, MD (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor-Investigator, Kami Maddocks, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-10052; NCI-2011-03293 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-11-01; First posted 2011-11-28 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — ibrutinib; Rituximab; Bendamustine Hydrochloride; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (enzyme inhibitor, chemo, monoclonal antibody) (Experimental): Patients receive BTK inhibitor PCI-32765 PO QD on days 1-28. Patients also receive rituximab IV on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may continue receiving BTK inhibitor PCI-32765 PO in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: BTK inhibitor PCI-32765; Biological: rituximab; Drug: bendamustine hydrochloride; Other: pharmacogenomic studies; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: BTK inhibitor PCI-32765 — Given PO
  Other Names: Bruton's tyrosine kinase inhibitor PCI-32765; PCI-32765
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of BTK inhibitor PCI-32765 when given together with rituximab and bendamustine hydrochloride in treating patients with recurrent non-Hodgkin lymphoma (NHL). BTK inhibitor PCI-32765 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving BTK inhibitor PCI-32765 together with rituximab and bendamustine hydrochloride may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify the specific toxicities and a recommended phase 2 dose of PCI-32765 (BTK inhibitor PCI-32765) orally (PO) in combination with rituximab and bendamustine (bendamustine hydrochloride) (i.e., "combination therapy") in patients with relapsed and refractory B-cell NHL.

SECONDARY OBJECTIVES:

I. Evaluate the activity of combined rituximab, bendamustine, and PCI-32765 in patients with relapsed and refractory B-cell NHL as measured by response rate and duration of response.

II. Identify potential marker(s) predictive of response to the combination therapy.

III. Correlate pharmacogenetic (PGx) findings with patient response and toxicity.

OUTLINE: This is a dose-escalation study of BTK inhibitor PCI-32765.

Patients receive BTK inhibitor PCI-32765 PO once daily (QD) on days 1-28. Patients also receive rituximab intravenously (IV) on day 1 and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients may continue receiving BTK inhibitor PCI-32765 PO in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 4 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell NHL of the following subtypes: follicular, marginal zone (nodal, splenic, or extranodal), Waldenstrom's macroglobulinemia, diffuse large B-cell (DLCL) or mantle cell lymphoma (MCL) according to 2008 World Health Organization (WHO) criteria that is relapsed or refractory after at least 1 prior therapy

  * Patients with DLCL must be relapsed or refractory after previous autologous stem cell transplant unless transplant is contraindicated
  * Patients with MCL, follicular lymphoma (FL), marginal zone lymphoma, or Waldenstrom's macroglobulinemia are eligible after >= 1 prior therapies; however, patients with MCL who are not eligible for stem cell transplant (due to age or other co-morbidities) or refuse up-front stem cell transplantation may receive study treatment as their first-line therapy
* Body weight >= 40 kg
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Agreement to use contraception during the study and for 30 days after the last dose of study drug if sexually active and able to bear children
* Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local patient privacy regulations)

Exclusion Criteria:

* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the patient has been disease free for at least 2 years or which will not limit survival to < 2 years (Note: these cases must be discussed with the Principal Investigator)
* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of PCI-32765 PO, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Any immunotherapy, chemotherapy, radiotherapy, or experimental therapy within 3 weeks before first dose of study drug (corticosteroids for disease-related symptoms allowed but require 1-week washout before study drug administration)
* Use of medications known to prolong QTc interval or that may be associated with Torsades de Pointes are prohibited within 7 days of starting study drug and during treatment
* Central nervous system (CNS) involvement by lymphoma
* Grade >= 2 toxicity (other than alopecia) related to prior anticancer therapy including radiation
* Known history of human immunodeficiency virus (HIV), active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV surface antigen positive), carriers of HBV (surface antigen and surface antibody negative, but HBV core antibody positive), or any uncontrolled active systemic infection
* Major surgery within 4 weeks before first dose of study drug
* Previous serious infusion reactions or hypersensitivity to rituximab or bendamustine not controlled or prevented by steroid pre-medication
* Creatinine > 2.0 mg/dL
* Total bilirubin > 1.5 x upper limit of normal (ULN) (unless due to Gilbert's disease)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 x ULN
* Absolute neutrophil count (ANC) < 1000/mm^3
* Platelets < 50,000/mm^3
* Lactating or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) as determined by the incidence of dose limiting toxicities (DLT) of BTK inhibitor PCI-32765 when given in combination with rituximab and bendamustine hydrochloride | during first course of therapy
  MTD is defined as the highest dose Level at which =< 1 of 6 patients experienced a DLT.

SECONDARY OUTCOMES:
Frequency, severity, and relatedness of adverse events | up to 30 days after last dose of treatment
  Laboratory shift tables containing counts and percentages will be prepared by treatment assignment, laboratory parameter, and time. Summary tables will be prepared for each laboratory parameter. Figures of changes in laboratory parameters over time will be generated.
Overall response rate | up to 24 months post treatment
  The point estimate of the rate will be calculated for the per protocol analysis set. The response rate 95% confidence interval estimates also will be derived. Association between the correlation markers and response will be explored using graphical and descriptive analysis.
Duration of response | up to 24 months post treatment
  From time measurement criteria are met for complete response(CR)or partial response(PR)until the first date that recurrent or progressive disease occurs. Median duration of overall response will be assessed with 95% confidence interval.
Identification of germinal center versus nongerminal center DLCL | screening or cycle 1 day 1 predose
  Determined by immunohistochemistry in patients with DLCL enrolled in the dose escalation portion of the study and in the DLCL expansion cohort.
Correlation of PGx with response and toxicity | screening or cycle 1 day 1 predose
  Data will be evaluated with pharmacokinetics and clinical outcomes to identify significant associations and potential PGx biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Kami Maddocks, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Maddocks K, Christian B, Jaglowski S, Flynn J, Jones JA, Porcu P, Wei L, Jenkins C, Lozanski G, Byrd JC, Blum KA. A phase 1/1b study of rituximab, bendamustine, and ibrutinib in patients with untreated and relapsed/refractory non-Hodgkin lymphoma. Blood. 2015 Jan 8;125(2):242-8. doi: 10.1182/blood-2014-08-597914. Epub 2014 Oct 29. PMID 25355819
- See also: Jamesline — http://cancer.osu.edu